CLINICAL TRIAL: NCT02542527
Title: C88- Pilot Study A Prospective Case Series for Evaluation of the Functionality of a Fluid Filled Single Breast Pump Applied on a Lactating Breast
Brief Title: Evaluation of the Functionality of a Fluid Filled Single Breast Pump
Acronym: C88
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MBF1504
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2015-10

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pumping with a fluid filled breast pump (Experimental): Participants pump (each breast 25 min) with the new fluid filled breast pump
  Interventions: Procedure: Fluid filled breast pump

INTERVENTIONS:
Procedure: Fluid filled breast pump — breast milk pumping with a fluid filled breast pump

SUMMARY:
This study is an early (during the product development process) feasibility study. It shall evaluate the device design concept with respect to device functionality of a new fluid filled breast pump in a small number of subjects.

ELIGIBILITY:
Inclusion criteria:

* Female over 18 years
* Participant has an established milk flow, general rule: approx. 50 ml per breast per pumping session
* The participant is pumping at least 2 times a week
* The participant is 1-6 months after giving birth (postpartum) at the day of data assessment
* The participant agrees to pump or feed the last time a minimum of 3 hours before the start of the pumping sessions
* The participant agrees that the pumped breast milk cannot be fed to her infant (will be disposed)
* The participant agrees to photograph and video record the breast and upper body (no face)
* The participant agrees to the presence of up to 3 men in the room during the pumping session

Exclusion criteria:

* Participant or their baby is dependent on life-sustaining electric devices (e.g. heart pacemaker, insulin pump, etc.)
* Participant has an medical condition of the breast
* Participant is allergic to plastics or silicone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Breast pump vacuum (mmHg) | Measured during a single 25 minute pumping session
  Vacuum will be continuously recorded during a single 25 Minute pumping session. The recorded units will be in mmHg. Each participants data will be assessed for the Minimum value, the Maximum value and the Mean value over 25 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Prime, PhD, Principal Investigator — Medela Switzerland
Locations (1):
- Medela AG, Baar, Canton of Zug, Switzerland